CLINICAL TRIAL: NCT07018063
Title: Efficacy and Safety of Neoadjuvant Nab-Paclitaxel Combined With Oxaliplatin, S-1, and Sintilimab in Patients With Locally Advanced Resectable Early-onset Gastric Cancer: A Phase II, Single-Arm, Open-Label Clinical Trial
Brief Title: Neoadjuvant Nab-Paclitaxel Plus Oxaliplatin, S-1, and Sintilimab in Early-Onset Resectable Gastric Cancer
Acronym: YOUNG-NEOS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: zhoujing (Other)
Responsible Party: Sponsor-Investigator, zhoujing, Chief Medical Oncologist, Department of Gastrointestinal Surgery, Peking University People's Hospital, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-EOGC-001
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Gastric (Cardia, Body) Cancer; Stomach Adenocarcinoma; Locally Advanced
Keywords: gastric cancer; Neoadjuvant therapy; Early-onset gastric cancer; Immunotherapy; Chemotherapy; Single-arm trial; Phase II trial; Perioperative treatment; China
MeSH Terms: conditions — Neoplasms; Stomach Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Oxaliplatin; S 1 (combination); sintilimab

STUDY DESIGN:
Intervention Model Description: All enrolled participants will receive the investigational treatment. No control group is included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant nab-SOX plus Sintilimab (Experimental): Patients will receive three 3-week cycles of neoadjuvant chemotherapy consisting of nab-paclitaxel 125 mg/m² IV on day 1, oxaliplatin 85 mg/m² IV on day 1, and S-1 80-120 mg/day orally on days 2-15, plus sintilimab 200 mg IV on day 1. D2 gastrectomy will be performed 3-6 weeks after neoadjuvant therapy.
  Interventions: Drug: nab-paclitaxel; Drug: oxaliplatin; Drug: S-1; Drug: sintilimab; Procedure: D2 Gastrectomy

INTERVENTIONS:
Drug: nab-paclitaxel — Nab-paclitaxel is administered as an intravenous (IV) infusion at a dose of 125 mg/m² on day 1 of each 3-week cycle, for a total of 3 cycles in the neoadjuvant (preoperative) setting.
Drug: oxaliplatin — Oxaliplatin is administered as an intravenous (IV) infusion at a dose of 85 mg/m² on day 1 of each 3-week cycle, for a total of 3 cycles in the neoadjuvant (preoperative) setting.
Drug: S-1 — S-1 is administered orally twice daily (BID) on days 2 to 15 of each 3-week cycle, for a total of 3 cycles. The dose is based on body surface area (BSA) as follows:
  BSA < 1.25 m²: 40 mg BID (total 80 mg/day); BSA 1.25-1.5 m²: 50 mg BID (total 100 mg/day); BSA > 1.5 m²: 60 mg BID (total 120 mg/day)
Drug: sintilimab — Sintilimab is administered as an intravenous (IV) infusion at a fixed dose of 200 mg on day 1 of each 3-week cycle, for a total of 3 cycles in the neoadjuvant (preoperative) setting.
Procedure: D2 Gastrectomy — Curative-intent D2 radical gastrectomy is performed 3 to 6 weeks after completion of neoadjuvant therapy. The procedure includes either proximal, distal or total gastrectomy depending on tumor location, with en bloc resection of the stomach and systematic D2 lymphadenectomy according to Japanese Gastric Cancer Association (JGCA) guidelines. D2 lymph node dissection involves removal of both perigastric (N1) and second-tier (N2) lymph nodes.

SUMMARY:
This study aims to evaluate the effectiveness and safety of a preoperative treatment (called neoadjuvant therapy) combining four drugs-nab-paclitaxel, oxaliplatin, S-1, and sintilimab-for patients with locally advanced, resectable early-onset gastric cancer (diagnosed at age 45 or younger).

All participants will receive this drug combination before undergoing surgery to remove the tumor. The goal is to shrink the tumor, increase the chance of complete surgical removal, and improve long-term outcomes.

This is a single-arm, open-label, phase II clinical trial, meaning all participants will receive the same treatment, and both doctors and patients will know what drugs are being used. The study is being conducted at Peking University People's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following inclusion criteria:
* Male or female, aged ≥16 and ≤45 years;
* Karnofsky performance score ≥70% or ECOG performance status 0-1;
* Histologically confirmed adenocarcinoma of the stomach or gastroesophageal junction (GEJ).
* For gastric body cancer: clinical stage cT3-T4a N+ M0;
* For GEJ cancer: clinical stage cT2-T4a N+ M0;
* For cT4b Nany M0 cases: location may be gastric body or GEJ.
* Staging is based on contrast-enhanced CT, MRI (if needed), and endoscopic ultrasonography (EUS) (if needed);
* Assessed as resectable after multidisciplinary team (MDT) discussion;
* Surgical evaluation confirms that D2 radical gastrectomy is feasible;
* Sufficient physical condition and organ function to tolerate major abdominal surgery;
* Baseline laboratory tests meet the following criteria:
* Hemoglobin ≥90 g/L
* Absolute neutrophil count (ANC) ≥1.5×10⁹/L
* Platelets ≥100×10⁹/L
* ALT and AST ≤2.5× upper limit of normal (ULN)
* Alkaline phosphatase (ALP) ≤2.5× ULN
* Total bilirubin <1.5× ULN
* Serum creatinine <1× ULN
* Serum albumin ≥30 g/L
* No severe comorbidities that may limit life expectancy to <3 years;
* Participant is willing and able to comply with the study protocol during the study period;
* Written informed consent must be signed before screening. Participants must understand their right to withdraw at any time without any loss of benefits;
* Willing to provide blood and tissue samples.

Exclusion Criteria:

* Participants meeting any of the following criteria will be excluded:
* Patients with HER-2 positive gastric cancer, as determined by immunohistochemistry (IHC) or fluorescence in situ hybridization (FISH);
* Patients with dMMR (deficient mismatch repair) or MSI-H (microsatellite instability-high) tumors, as determined by IHC;
* Pregnant or breastfeeding women;
* Prior treatment for gastric cancer with cytotoxic chemotherapy, radiotherapy, or immunotherapy;
* History of other malignancies within the past 5 years;
* Active autoimmune diseases, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, myasthenia gravis;
* Active inflammatory bowel diseases, such as Crohn's disease or ulcerative colitis;
* Currently receiving systemic corticosteroids or other immunosuppressive therapy;
* Prior organ transplantation or use of anti-rejection medications;
* Active tuberculosis, HIV infection, or severe active hepatitis B or C;
* History of uncontrolled epilepsy, central nervous system disorders, or psychiatric illnesses that, in the investigator's judgment, may interfere with informed consent or compliance with oral medication;
* Clinically significant (active) cardiac diseases, including symptomatic coronary artery disease, NYHA class II or above congestive heart failure , severe arrhythmias requiring medical intervention, or myocardial infarction within the past 12 months;
* Presence of upper gastrointestinal obstruction that may impair the oral intake or absorption of S-1;
* Severe uncontrolled recurrent infections or other uncontrolled serious comorbidities;
* Use of any investigational drugs within 4 weeks prior to study enrollment.

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate after neoadjuvant therapy | At the time of surgery, approximately 13-16 weeks from the start of neoadjuvant therapy
  Pathological complete response (pCR) is defined as the absence of residual invasive tumor cells in the resected stomach and lymph nodes (ypT0N0), as assessed by centralized pathological review following D2 radical gastrectomy.

SECONDARY OUTCOMES:
R0 resection rate after neoadjuvant therapy and surgery | At the time of surgery, approximately 13-16 weeks from the start of treatment
  The proportion of patients achieving R0 resection, defined as complete macroscopic and microscopic tumor removal with negative margins.
Major pathological response (MPR) rate based on Becker tumor regression grade | At the time of surgery, approximately 13-16 weeks from the start of treatment
  The proportion of patients with residual tumor cells ≤10% in the primary tumor bed, corresponding to Becker TRG 1a and 1b categories, assessed by pathological review.
3-year disease-free survival (DFS) | Up to 36 months after surgery
  DFS is defined as the time from informed consent to the first occurrence of tumor recurrence, metastasis, or death from any cause.
3-year overall survival (OS) | Up to 36 months after surgery
  OS is defined as the time from informed consent to death from any cause. Censoring will occur at the last follow-up for event-free patients.
Incidence of treatment-related grade 3 or higher adverse events | From initiation of treatment to surgery, approximately 12-15 weeks
  Frequency and types of grade 3 or higher adverse events as defined by NCI CTCAE v5.0, recorded during neoadjuvant therapy to evaluate treatment safety.
Incidence of major postoperative complications | From surgery until hospital discharge or 30 days postoperatively, whichever is longer
  Postoperative complications will be recorded and classified using the Clavien-Dindo classification system, including but not limited to anastomotic leakage, surgical site infection, and postoperative bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: JING ZHOU, M.D., Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices), will be shared with researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available beginning 6 months after publication and ending 5 years after publication.
Access Criteria: Researchers requesting data sharing should send their research proposals to xuesongzhao@bjmu.edu.cn. Access to the data will require consultation with the principal investigator and the signing of a data use agreement.

REFERENCES:
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Becker K, Mueller JD, Schulmacher C, Ott K, Fink U, Busch R, Bottcher K, Siewert JR, Hofler H. Histomorphology and grading of regression in gastric carcinoma treated with neoadjuvant chemotherapy. Cancer. 2003 Oct 1;98(7):1521-30. doi: 10.1002/cncr.11660. PMID 14508841
- [Background] Watson S, de la Fouchardiere C, Kim S, Cohen R, Bachet JB, Tournigand C, Ferraz JM, Lefevre M, Colin D, Svrcek M, Meurisse A, Louvet C. Oxaliplatin, 5-Fluorouracil and Nab-paclitaxel as perioperative regimen in patients with resectable gastric adenocarcinoma: A GERCOR phase II study (FOXAGAST). Eur J Cancer. 2019 Jan;107:46-52. doi: 10.1016/j.ejca.2018.11.006. Epub 2018 Dec 7. PMID 30529902
- [Background] Shitara K, Takashima A, Fujitani K, Koeda K, Hara H, Nakayama N, Hironaka S, Nishikawa K, Makari Y, Amagai K, Ueda S, Yoshida K, Shimodaira H, Nishina T, Tsuda M, Kurokawa Y, Tamura T, Sasaki Y, Morita S, Koizumi W. Nab-paclitaxel versus solvent-based paclitaxel in patients with previously treated advanced gastric cancer (ABSOLUTE): an open-label, randomised, non-inferiority, phase 3 trial. Lancet Gastroenterol Hepatol. 2017 Apr;2(4):277-287. doi: 10.1016/S2468-1253(16)30219-9. Epub 2017 Jan 19. PMID 28404157
- [Background] Zhang C, Tang R, Zhu H, Ge X, Wang Y, Wang X, Miao L. Comparison of treatment strategies and survival of early-onset gastric cancer: a population-based study. Sci Rep. 2022 Apr 15;12(1):6288. doi: 10.1038/s41598-022-10156-5. PMID 35428811
- [Background] Liu L, Lin J, Zhao J, Yan P. Analysis of clinicopathologic characteristics and prognosis of gastric cancer in patients <40 years. Medicine (Baltimore). 2023 Aug 25;102(34):e34635. doi: 10.1097/MD.0000000000034635. PMID 37653814
- [Background] Liu JD, Ye BT, Fu M, Zhang Q, Chen H, Sun J, Cai TY, Wang ZM, He HY, Zhao JJ, Li HJ, Wang XF, Sun YH. [Clinicopathological and molecular diagnostic features of early-onset gastric cancer: a study based on data from a single-center dedicated gastric cancer database]. Zhonghua Wei Chang Wai Ke Za Zhi. 2023 Oct 25;26(10):963-967. doi: 10.3760/cma.j.cn441530-20230603-00190. Chinese. PMID 37849267
- [Background] Pocurull A, Herrera-Pariente C, Carballal S, Llach J, Sanchez A, Carot L, Botargues JM, Cuatrecasas M, Ocana T, Balaguer F, Bujanda L, Moreira L. Clinical, Molecular and Genetic Characteristics of Early Onset Gastric Cancer: Analysis of a Large Multicenter Study. Cancers (Basel). 2021 Jun 23;13(13):3132. doi: 10.3390/cancers13133132. PMID 34201547
- [Background] Rompen IF, Nienhuser H, Crnovrsanin N, Musa J, Haag GM, Longerich T, Fiedler T, Muller-Stich BP, Sisic L, Billeter AT. Clinical Characteristics and Oncological Outcomes of Surgically Treated Early-Onset Gastric Adenocarcinoma - a Retrospective Cohort Study. J Cancer. 2023 May 21;14(9):1470-1478. doi: 10.7150/jca.82876. eCollection 2023. PMID 37325055
- [Background] Qu X, Zhao X, Liu Y, Wang N, Zhang L, Zhu X, Dong Q, Liu J, Shi Y. The clinicopathological characteristics of early-onset gastric cancer and its evolutionary trends: a retrospective study. Am J Cancer Res. 2022 Jun 15;12(6):2757-2769. eCollection 2022. PMID 35812046
- [Background] Ning FL, Zhang NN, Zhao ZM, Du WY, Zeng YJ, Abe M, Pei JP, Zhang CD. Global, Regional, and National Burdens with Temporal Trends of Early-, Intermediate-, and Later-Onset Gastric Cancer from 1990 to 2019 and Predictions up to 2035. Cancers (Basel). 2022 Nov 3;14(21):5417. doi: 10.3390/cancers14215417. PMID 36358835
- [Background] Lumish MA, Walch H, Maron SB, Chatila W, Kemel Y, Maio A, Ku GY, Ilson DH, Won E, Li J, Joshi SS, Gu P, Schattner MA, Laszkowska M, Gerdes H, Jones DR, Sihag S, Coit DG, Tang LH, Strong VE, Molena D, Stadler ZK, Schultz N, Janjigian YY, Cercek A. Clinical and molecular characteristics of early-onset vs average-onset esophagogastric cancer. J Natl Cancer Inst. 2024 Feb 8;116(2):299-308. doi: 10.1093/jnci/djad186. PMID 37699004